CLINICAL TRIAL: NCT05047809
Title: The Evaluation of Treatment of Leprosy Wounds With Traditional Chinese Herbal Medicine Complex "Jingchuang Ointment"
Brief Title: The Effect of "Jinchuang Ointment" (JCO) on the Treatment of Wounds in Patients With Hansen's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo-Sheng Sanatorium (Other Government)
Responsible Party: Principal Investigator, Hsu Wei Hung, Director of chinese medicine, Lo-Sheng Sanatorium
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYGH110014
Record Dates: First submitted 2021-08-25; First posted 2021-09-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Leprosy; Hansen's Disease; Wounds
Keywords: Leprosy; Hansen's disease (HD); Jinchuang Ointment (JCO); wounds; anti-inflammation
MeSH Terms: conditions — Leprosy; Wounds and Injuries | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Jingchuang Ointment"(JCO) group (Experimental): Ulcers were treated in this study using the four-step wound care guidelines, observation, rinsing, cleaning, and dressing, published by the Taiwan Food and Drug Administration. Besides, JCO was applied once a day on the wounds, last 3 months.
  "Jingchuang Ointment" (JCO) is made by Chuang Song Zong Pharmaceutical Co., Ltd. (Taiwan)
  Interventions: Other: "Jingchuang Ointment"(JCO)
- Regular treatment group (Other): Ulcers were treated in this study using the four-step wound care guidelines, observation, rinsing, cleaning, and dressing, published by the Taiwan Food and Drug Administration.
  Interventions: Other: Regular Treatment

INTERVENTIONS:
Other: "Jingchuang Ointment"(JCO) — Applied once a day on the wounds
  Other Names: Chuang Song Zong Pharmaceutical Co., Ltd. (Taiwan)
  Arms: "Jingchuang Ointment"(JCO) group
Other: Regular Treatment — Do not use the "Jingchuang Ointment"(JCO), as the regular treatment as usual.
  Arms: Regular treatment group

SUMMARY:
This study aimed to evaluate the effect of a Chinese herb complex "Jinchuang ointment" (JCO) on the treatment of chronic nonhealing wounds in patients with Hansen's disease and its mechanism.

DETAILED DESCRIPTION:
20 patients who were hospitalized at Lo-Sheng Sanatorium, Ministry of Health and Welfare, were recruited. Ulcers were treated in this study using the four-step wound care guidelines, observation, rinsing, cleaning, and dressing, published by the Taiwan Food and Drug Administration. Besides, JCO was applied once a day on the wounds.

Basic data of each case were collected, and a monthly wound record was used to follow the condition of the wound healing of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Hanson's patients
* Meet the definition of chronic wound

Exclusion Criteria:

* Kidney disease
* Parathyroid disease
* Malignant tumors.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-07 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
The size of wound area | Changes in wound size in 3 months
  Length times width

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Hung Hsu, Principal Investigator — Lo-Sheng Sanatorium
Locations (1):
- Lo-Sheng Sanatorium, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-05-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT05047809/ICF_000.pdf